CLINICAL TRIAL: NCT02405741
Title: Does Hyperbaric Chamber Improve the Functionality and Symptoms Related to Central Retinal Vein Occlusion (CRVO)?
Brief Title: Hyperbaric Chamber for Central Retinal Vein Occlusion (CRVO) Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Dr. Shai Efrati, Assaf-Harofeh Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 238/14
Record Dates: First submitted 2015-03-23; First posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Central Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Hyperbaric chamber treatment

SUMMARY:
Hyperbaric chamber treatment assists in increasing the amount of oxygen in the plasma and in the tissues and has been proven to be beneficial in treating different ischemic wounds, and acute retinal artery occlusion (ARAO) but its effect hasn't been tested in CRVO patients yet.

DETAILED DESCRIPTION:
Trial protocol V2.0 - Hyperbaric chamber treatment to CRVO patients

Assaf HaRofe Medical Center - Zerifin, Israel

Purpose: To determine whether hyperbaric chamber treatment improves the functionality and symptoms related to CRVO

Introduction:

Central Retinal Vein Occlusion (CRVO) has profound effects on retinal circulation. As this vein collects the entire venous outflow from the retina, retinal perfusion is greatly impaired when it occludes. Even though, as compensation, the collateral outflow is expanded but nevertheless there is an increase in retinal venous pressure, venous dilation, retinal hemorrhage and retinal edema.

Reduction of blood flow leads to retinal hypoxia and upregulation of vascular endothelial growth factor (VGEF )

In CRVO there is a variable degree of capillary nonperfusion visible on fluorescein angiography (FA) which is divided into "ischemic" and "non ischemic" depending on the size of the area of non perfusion on FA.

Possible complications of CRVO include chronic cystoid macular edema (CME), neovascularization of retina, neovascular glaucoma and vitreous hemorrhage. These complications are serious, sight threatening, and require prolonged treatment.

Current therapy of CRVO requires different treatment modalities depending on the complication.

Neovascularization is treated mainly by laser photocoagulation (PRP - pan retinal photocoagulation) and VEGF inhibitors. Photocoagulation is based on lowering the oxygen consumption of peripheral retina.

Macular edema is treated with anti VEGF and/or steroidal injections. Most patients require continuous monthly injections which may last for years in order to dehydrate their macula.

Recent clinical trials such as CRUISE and BRAVO have shown that the immediate monthly injections of anti VEGF (Ranibizumab) during the first 6 months and then later as needed decreased substantially the time to achieve visual acuity gain following CRVO5. In BRAVO trial the cumulative proportion of patients who had gained 15 letters or more from baseline by 12 month (from CRVO incidence) was 50% (sham), 68% (ranibizumab 0.3 mg), and 71% (ranibizumab 0.5 mg) and in CRUISE trial 42%, 61%, and 66%, respectively.

Another trial which evaluated the effect of anti VEGF was the COPERNICUS trial in which patients with CRVO received intravitreal aflibercept injection every 4 weeks up to 6 months following the CRVO. The control group received sham injections and the proportion of patients gaining ≥ 15 letters was 56.1% versus 12.3% (P<0.001) at week 24. Improved reduction in central retinal thickness and increased vitreous hemorrhage as the major side effect (up to 6.8%) was also evident in patients treated with aflibercept.

Although effective, these anti VEGF injections expose the patient to many possible side effects including sub conjunctival hemorrhage and transient hypertension at the mild end of the spectrum or endophthalmitis and lens injury at the severe end.

An alternative treatment is the use of steroids such as dexamethasone intravitreal implant (Ozurdex). However, this treatment may induce side effects such as increased ocular pressure, cataract, allergy, conjunctival hemorrhage and eye pain.

Hypoxic induction of cytokines, such as VEGF, play a central role in CRVO and its consequences such as retinal edema and iris neovascularization.

Hyperbaric chamber has the potential to increase oxygen perfusion and perhaps decrease retinal hypoxia, thereby decreasing the induction of cytokines and improving retinal functionality.

The investigators' broad experience in hyperbaric chamber treatment reveals that it is a rather benign treatment compared to the alternatives where the most relevant side effect in eligible patients is usually ear barotrauma.

Investigative Device:

Hyperbaric chamber assists in increasing the amount of oxygen in the plasma and in the tissues and has been proven to be beneficial in treating different ischemic wounds, and acute retinal artery occlusion (ARAO) but its effect hasn't been tested in CRVO patients yet.

Methods:

Patients with chronic CRVO who are receiving monthly injections of Bevacizumab treatment for at least 12 months will be recruited. Upon recruitment each patient will undergo a screening Ophthalmologic examination including visual acuity, refraction and OCT. This will be followed by a series of 40 daily hyperbaric chamber treatments. A repeated ophthalmic examination will be done after 20 and 40 hyperbaric sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18-80 years with a documented CRVO who treated by Avastin for more than 12 months.
2. Patients who signed an informed consent form

Exclusion Criteria:

1. Patients with Carotid stenosis of more than 70%
2. Anemia of < 10mg/Dl
3. Patients with chest X ray pathology which cannot be admitted to hyperbaric chamber treatment.
4. Patients with claustrophobia or that cannot decompress properly.
5. Patients with any malignant disease
6. Patients with inability to sign informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Optical Coherence Tomography Measurements of the Retina | up to 40 treatments (expected average of 8 weeks)
  This is a non-contact medical imaging technology similar to ultrasound and MRI. With OCT, reflected light is used to produce detailed cross-sectional and 3D images of the eye.

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofe MC, Ẕerifin, Israel